CLINICAL TRIAL: NCT05715333
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Immunogenicity of CM326 Injection in Healthy Subjects
Brief Title: Study of CM326 Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM326-100003
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2023-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): CM326 220 mg/2 mL or matched placebo, subcutaneous at low dose
  Interventions: Biological: CM326; Other: Placebo
- Group 2 (Experimental): CM326 220mg/2 mL or matched placebo, subcutaneous at medium dose
  Interventions: Biological: CM326; Other: Placebo
- Group 3 (Experimental): CM326 220mg/2mL or matched placebo, subcutaneous at high dose
  Interventions: Biological: CM326; Other: Placebo
- Group 4 (Experimental): CM326 220mg/2mL or matched placebo, subcutaneous at medium dose
  Interventions: Biological: CM326; Other: Placebo

INTERVENTIONS:
Biological: CM326 — CM326 Injection
Other: Placebo — Subcutaneous injection

SUMMARY:
This study is a single-center, randomized, double-blind, placebo-controlled, dose-increasing phase I clinical study.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerance, pharmacokinetics and immunogenicity of single and multiple subcutaneous administration of CM326 at different doses in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤ 65 years, healthy male.
* With normal or abnormal laboratory test results without clinical significanceat screening period and baseline.
* Subjects can communicate well with investigators and comply with protocol requirements.

Exclusion Criteria:

* Any live attenuated vaccine is planned to be inoculated 30 days before administration or during the study period.
* Major surgery is planned during the study period.
* The average daily smoking volume is more than 5 cigarettes within 3 months before screening.
* Within 12 weeks before administration, blood loss from voluntary blood donation or any attempt to visit is greater than 400 mL.
* There are any reasons that the investigator believes will prevent the subject from participating in the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Emergency adverse events during treatment | Up to week 12
  By assessing the number and severity of adverse events during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Hou, Principal Investigator — Peking University Care Luzhong Hospital; Hong Wang, Principal Investigator — Peking University Care Luzhong Hospital
Locations (1):
- PKUCare Luzhong Hospital, Zibo, China

REFERENCES:
- [Derived] Di Y, Yang L, Zhou J, Zhang L, Huang Y, Jia Y, Yan H, Chen L, Hou Q, Chen B, Luo Z, Hou J. Translational Investigation of CM326 from Preclinical Studies to Randomized Phase I Clinical Trials in Healthy Adults. BioDrugs. 2025 May;39(3):487-498. doi: 10.1007/s40259-025-00714-4. Epub 2025 Apr 4. PMID 40185989